CLINICAL TRIAL: NCT02507973
Title: Study of APRV and ICP in Patients With Severe Traumatic Brain Injury
Brief Title: Study of Airway Pressure Release Ventilation and Intracranial Pressure in Patients With Severe Traumatic Brain Injury
Status: Terminated | Type: Observational
Why Stopped: Unable to successfully recruit patients for study.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deborah Stein, Medical Director, Neurotrauma Critical Care; Chief, Section of Trauma Critical Care, R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Other Study IDs: HP-00063355
Record Dates: First submitted 2015-07-17; First posted 2015-07-24 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Injury, Brain, Traumatic; Traumatic Brain Injury
Keywords: Mechanical Ventilation; Intracranial Pressure; Airway Pressure Release Ventilation
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Airway Pressure Release Ventilation:APRV: Each participant will serve as his/her own control using our observational crossover study comparing the effects of Airway Pressure Release Ventilation and Low Tidal Volume Ventilation on patient intracranial pressure and hemodynamic values.
  Interventions: Other: Airway Pressure Release Ventilation
- Low Tidal Volume Ventilation:LOTV: Each participant will serve as his/her own control using our observational crossover study comparing the effects of Airway Pressure Release Ventilation and LOTV on patient intracranial pressure and hemodynamic values.
  Interventions: Other: Low Tidal Volume Ventilation

INTERVENTIONS:
Other: Airway Pressure Release Ventilation — Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that switches between high (PHigh) and low (PLow) continuous positive airway pressure while allowing spontaneous breathing at both phases. Alveolar recruitment and oxygenation occur during PHigh whereas ventilation occurs during brief releases to PLow.
  Other Names: APRV
  Groups: Airway Pressure Release Ventilation:APRV
Other: Low Tidal Volume Ventilation — After enrollment and collection of baseline Intracranial pressure and hemodynamic status for 30 minutes the participants will undergo low tidal volume mechanical ventilation (LOTV), serving as a control mode of ventilation. LOTV is most commonly used for trauma patients with lung injury. LOTV provides oxygen in smaller amounts, without overstretching the lungs
  Other Names: LOTV
  Groups: Low Tidal Volume Ventilation:LOTV

SUMMARY:
The investigators will conduct an observational crossover study. The investigators aim to recruit 50 participants with severe Traumatic Brain Injury (TBI) requiring intracranial pressure (ICP) monitoring during their stay at the Neuro Trauma ICU at the R Adams Cowley Shock Trauma Center.

Overall, participants will be monitored, on average, for approximately 6-8 hours during the study period. The investigators do not anticipate the need for prolonged monitoring during the duration of their hospital stay or post hospital period.

DETAILED DESCRIPTION:
Each participant at admission will initially receive a primary mode of mechanical ventilation as determined by the attending trauma intensivists. 12-18 hours after recruitment, continuous monitoring of participants' ICP and hemodynamic status will commence to collect participants' baseline data for 30 minutes.

Participants will then undergo low tidal volume mechanical ventilation (LOTV), serving as a control mode of ventilation, for 2 hours prior to switching back to the primary mode of ventilation for 30 minutes. Next, patients will be placed on Airway Pressure Release Ventilation (APRV) for 2 hours. While receiving APRV, participants Intracranial pressure and hemodynamic status will be continuously monitored and recorded for comparison and analysis. After 2 hours of APRV, patients will be switched back to their previous mode of ventilation and more data collected for another 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial Pressure Monitoring device present
* Mechanically Ventilated
* Clinically Stable as determined by the Critical Care attending

Exclusion Criteria:

* Age <14
* Prisoners
* Initial Mode of ventilation is APRV
* Provider's Judgement
* Pregnant

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with intracranial pressure monitor requiring mechanical ventilation support will be eligible for enrollment in the study
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Stein, MD, MPH, Principal Investigator — Professor, Department of Surgery
Locations (1):
- RA Cowley Shock Trauma Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosio A. A theoretical study of new types of valve shunts for cerebrospinal fluid. ASAIO Trans. 1991 Jul-Sep;37(3):M289-90. PMID 1751154
- [Background] Chesnut RM, Marshall SB, Piek J, Blunt BA, Klauber MR, Marshall LF. Early and late systemic hypotension as a frequent and fundamental source of cerebral ischemia following severe brain injury in the Traumatic Coma Data Bank. Acta Neurochir Suppl (Wien). 1993;59:121-5. doi: 10.1007/978-3-7091-9302-0_21. PMID 8310858
- [Background] Fearnside MR, Cook RJ, McDougall P, McNeil RJ. The Westmead Head Injury Project outcome in severe head injury. A comparative analysis of pre-hospital, clinical and CT variables. Br J Neurosurg. 1993;7(3):267-79. doi: 10.3109/02688699309023809. PMID 8338647
- [Background] Schreiber MA, Aoki N, Scott BG, Beck JR. Determinants of mortality in patients with severe blunt head injury. Arch Surg. 2002 Mar;137(3):285-90. doi: 10.1001/archsurg.137.3.285. PMID 11888450
- [Background] Jones PA, Andrews PJ, Midgley S, Anderson SI, Piper IR, Tocher JL, Housley AM, Corrie JA, Slattery J, Dearden NM, et al. Measuring the burden of secondary insults in head-injured patients during intensive care. J Neurosurg Anesthesiol. 1994 Jan;6(1):4-14. PMID 8298263
- [Background] Stocchetti N, Furlan A, Volta F. Hypoxemia and arterial hypotension at the accident scene in head injury. J Trauma. 1996 May;40(5):764-7. doi: 10.1097/00005373-199605000-00014. PMID 8614077
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. VIII. Intracranial pressure thresholds. J Neurotrauma. 2007;24 Suppl 1:S55-8. doi: 10.1089/neu.2007.9988. No abstract available. PMID 17511546
- [Background] Marshall LF, Smith RW, Shapiro HM. The outcome with aggressive treatment in severe head injuries. Part I: the significance of intracranial pressure monitoring. J Neurosurg. 1979 Jan;50(1):20-5. doi: 10.3171/jns.1979.50.1.0020. No abstract available. PMID 758374
- [Background] Saul TG, Ducker TB. Intracranial pressure monitoring in patients with severe head injury. Am Surg. 1982 Sep;48(9):477-80. PMID 7125382
- [Background] Narayan RK, Kishore PR, Becker DP, Ward JD, Enas GG, Greenberg RP, Domingues Da Silva A, Lipper MH, Choi SC, Mayhall CG, Lutz HA 3rd, Young HF. Intracranial pressure: to monitor or not to monitor? A review of our experience with severe head injury. J Neurosurg. 1982 May;56(5):650-9. doi: 10.3171/jns.1982.56.5.0650. No abstract available. PMID 7069477
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. XI. Anesthetics, analgesics, and sedatives. J Neurotrauma. 2007;24 Suppl 1:S71-6. doi: 10.1089/neu.2007.9985. No abstract available. PMID 17511550
- [Background] Nyquist P, Stevens RD, Mirski MA. Neurologic injury and mechanical ventilation. Neurocrit Care. 2008;9(3):400-8. doi: 10.1007/s12028-008-9130-7. Epub 2008 Aug 12. PMID 18696268
- [Background] Stevens RD, Lazaridis C, Chalela JA. The role of mechanical ventilation in acute brain injury. Neurol Clin. 2008 May;26(2):543-63, x. doi: 10.1016/j.ncl.2008.03.014. PMID 18514826
- [Background] Dries DJ, Marini JJ. Airway pressure release ventilation. J Burn Care Res. 2009 Nov-Dec;30(6):929-36. doi: 10.1097/BCR.0b013e3181bfb84c. No abstract available. PMID 19826261
- [Background] Habashi NM. Other approaches to open-lung ventilation: airway pressure release ventilation. Crit Care Med. 2005 Mar;33(3 Suppl):S228-40. doi: 10.1097/01.ccm.0000155920.11893.37. PMID 15753733
- [Background] Dart BW 4th, Maxwell RA, Richart CM, Brooks DK, Ciraulo DL, Barker DE, Burns RP. Preliminary experience with airway pressure release ventilation in a trauma/surgical intensive care unit. J Trauma. 2005 Jul;59(1):71-6. doi: 10.1097/00005373-200507000-00010. PMID 16096541
- [Background] Maung AA, Luckianow G, Kaplan LJ. Lessons learned from airway pressure release ventilation. J Trauma Acute Care Surg. 2012 Mar;72(3):624-8. doi: 10.1097/TA.0b013e318247668f. PMID 22491545
- [Background] Maxwell RA, Green JM, Waldrop J, Dart BW, Smith PW, Brooks D, Lewis PL, Barker DE. A randomized prospective trial of airway pressure release ventilation and low tidal volume ventilation in adult trauma patients with acute respiratory failure. J Trauma. 2010 Sep;69(3):501-10; discussion 511. doi: 10.1097/TA.0b013e3181e75961. PMID 20838119
- [Background] Andrews PL, Shiber JR, Jaruga-Killeen E, Roy S, Sadowitz B, O'Toole RV, Gatto LA, Nieman GF, Scalea T, Habashi NM. Early application of airway pressure release ventilation may reduce mortality in high-risk trauma patients: a systematic review of observational trauma ARDS literature. J Trauma Acute Care Surg. 2013 Oct;75(4):635-41. doi: 10.1097/TA.0b013e31829d3504. PMID 24064877
- [Background] Nemer SN, Caldeira JB, Azeredo LM, Garcia JM, Silva RT, Prado D, Santos RG, Guimaraes BS, Ramos RA, Noe RA, Souza PC. Alveolar recruitment maneuver in patients with subarachnoid hemorrhage and acute respiratory distress syndrome: a comparison of 2 approaches. J Crit Care. 2011 Feb;26(1):22-7. doi: 10.1016/j.jcrc.2010.04.015. Epub 2010 Jun 19. PMID 20646904
- [Background] Marik PE, Young A, Sibole S, Levitov A. The effect of APRV ventilation on ICP and cerebral hemodynamics. Neurocrit Care. 2012 Oct;17(2):219-23. doi: 10.1007/s12028-012-9739-4. PMID 22829002
- [Background] Kreyer S, Putensen C, Berg A, Soehle M, Muders T, Wrigge H, Zinserling J, Hering R. Effects of spontaneous breathing during airway pressure release ventilation on cerebral and spinal cord perfusion in experimental acute lung injury. J Neurosurg Anesthesiol. 2010 Oct;22(4):323-9. doi: 10.1097/ANA.0b013e3181e775f1. PMID 20622682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 patients were screened for eligibility between July 2015 and April 2018 at University of Maryland, Baltimore.
Pre-assignment Details: 8 of 200 patients were randomized. The other patients were excluded as they did not meet the eligibility criteria.
Groups:
- LOTV, Then APRV: Participants first were maintained on Low Tidal Volume Ventilation for two hours. Then there was a washout period of 30 minutes. After this washout period, they were maintained on Airway Pressure Release Ventilation for two hours.
  Each participant will serve as his/her own control using our observational crossover study comparing the effects of Airway Pressure Release Ventilation and Low Tidal Volume Ventilation on patient intracranial pressure and hemodynamic values.
  Airway Pressure Release Ventilation: Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that switches between high (PHigh) and low (PLow) continuous positive airway pressure while allowing spontaneous breathing at both phases. Alveolar recruitment and oxygenation occur during PHigh whereas ventilation occurs during brief releases to PLow.
Period: Overall Study
Arm/Group | LOTV, Then APRV
Started | 8
Completed | 7
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Participants first were maintained on Low Tidal Volume Ventilation for two hours. Then there was a washout period of 30 minutes. After this washout period, they were maintained on Airway Pressure Release Ventilation for two hours.
Groups:
- LOTV Then APRV: Participants first were maintained on Low Tidal Volume Ventilation for two hours. Then there was a washout period of 30 minutes. After this washout period, they were maintained on Airway Pressure Release Ventilation for two hours.
  Each participant will serve as his/her own control using our observational crossover study comparing the effects of Airway Pressure Release Ventilation and Low Tidal Volume Ventilation on patient intracranial pressure and hemodynamic values.
  Airway Pressure Release Ventilation: Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that switches between high (PHigh) and low (PLow) continuous positive airway pressure while allowing spontaneous breathing at both phases. Alveolar recruitment and oxygenation occur during PHigh whereas ventilation occurs during brief releases to PLow.
Arm/Group | LOTV Then APRV
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Patients Not Initially on APRV [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Pressure
Description: We aim to evaluate the patients during the two modes of ventilation (LTOV and APRV) to determine if there are significant differences in their ICP based on ventilation mode.
Time Frame: On average, 24 hours for each patient
Population: Access to original intracranial pressure data lost and cannot be summarized
  No data was analyzed to report.
Groups:
- LOTV; APRV: Participants first were maintained on Low Tidal Volume Ventilation for two hours. Then there was a washout period of 30 minutes. After this washout period, they were maintained on Airway Pressure Release Ventilation for two hours.
  Each participant will serve as his/her own control using our observational crossover study comparing the effects of Airway Pressure Release Ventilation and Low Tidal Volume Ventilation on patient intracranial pressure and hemodynamic values.
  Airway Pressure Release Ventilation: Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that switches between high (PHigh) and low (PLow) continuous positive airway pressure while allowing spontaneous breathing at both phases. Alveolar recruitment and oxygenation occur during PHigh whereas ventilation occurs during brief releases to PLow.
Arm/Group | LOTV | APRV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- LOTV; APRV: All Participants first were maintained on Low Tidal Volume Ventilation for two hours. Then there was a washout period of 30 minutes. After this washout period, they were maintained on Airway Pressure Release Ventilation for two hours.
  Each participant will serve as his/her own control using our observational crossover study comparing the effects of Airway Pressure Release Ventilation and Low Tidal Volume Ventilation on patient intracranial pressure and hemodynamic values.
  Airway Pressure Release Ventilation: Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that switches between high (PHigh) and low (PLow) continuous positive airway pressure while allowing spontaneous breathing at both phases. Alveolar recruitment and oxygenation occur during PHigh whereas ventilation occurs during brief releases to PLow.
  Patient's volume statuses and cardiac functions were assessed during the study period
  No data was analyzed to report.
Arm/Group | LOTV | APRV
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LOTV (N=8) | APRV (N=8)
Increased systolic blood pressure (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — One patient enrolled in the trial had a spike in systolic blood pressure to just above 300 mmHg when switched to APRV. The trial immediately terminated in this patient, and the systolic blood pressure returned to within normal limits.

LIMITATIONS AND CAVEATS:
This study was limited by poor patient enrollment. Thus, sufficient data was not collected for true analysis. Furthermore, access to LTOV and APRV intracranial pressure data lost and can not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT02507973/Prot_SAP_000.pdf